CLINICAL TRIAL: NCT00499876
Title: The Effect of Malaria on Disease Progression of HIV/AIDS in Kumasi, Ghana
Brief Title: The Effect of Malaria on Disease Progression of HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Noguchi Memorial Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: REG_9; KATH_GMP_1
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: HIV Infections; Malaria
Keywords: Human immune deficiency virus; Acquired immune deficiency syndrome; malaria; mefloquine; prophylaxis; HIV/AIDS; Treatment Naive
MeSH Terms: conditions — HIV Infections; Malaria; Acquired Immunodeficiency Syndrome | interventions — Mefloquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: mefloquine
- B (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: mefloquine — 250mg weekly PO for 6 months
  Arms: A
Other: placebo — 1 tablet weekly PO for 6 months
  Arms: B

SUMMARY:
The purpose of this study is to find out whether malaria affects how HIV/AIDS disease progresses in an infected patient, and to determine the effect of reducing malaria infection on HIV disease progression in Kumasi

DETAILED DESCRIPTION:
Malaria and HIV are among the most prevalent infectious diseases in sub-Saharan Africa and are major causes of morbidity and mortality in the sub region. Because of the wide-spread geographical overlap in HIV and malaria, the probability for co-infections and the potential for interactions between the two diseases are high. Even modest interactions may have substantial impact in populations.

It is now clear that there are interactions between the two infections. HIV associated immunosuppression erodes the malaria acquired immunity of the HIV patients. The risk of parasitaemia, high parasite density and malarial fever increases with decreasing CD4 T cell counts and increasing viral load of HIV patients. Plasmodium falciparum has been shown to stimulate HIV replication through the production of cytokines (including interleukin 6 and tumor necrosing factor α (TNF-α)) by activated lymphocytes. Malaria treatment in HIV patients with malaria resulted in significant reduction of the median HIV viral load concentration.

Although it is now clear that malaria causes transient rises in HIV-1 viral loads, could repeated episodes of malaria in areas of intense transmission lead to a cumulative effect on viral load and accelerate decline in CD4 counts thereby accelerating HIV disease progression? If so, could the decline in CD4 count in individuals who have not yet started on anti-retroviral drugs be slowed down by intermittent malaria treatment?

A controlled interventional study with mefloquine as malaria prophylaxis for 6 months will be used in HIV/AIDS patients who are not already on ARTs in KATH, and malaria parasitaemia and density, HIV viral load and CD4 cell count will be monitored in both arms.

Comparison: Malaria parasitaemia and density, HIV viral loads and CD4 cell counts will be compared between the intervention group and the control groups to determine the effect o malaria and malaria prophylaxis on HIV disease progression

ELIGIBILITY:
Inclusion Criteria:

* Adult HIV patients attending the Komfo Anokye Teaching Hospital (KATH) HIV clinic who do not yet fulfil the criteria for ARTs. This includes a CD 4 cell count of ≥ 300x106/l and World Health Organisation HIV stage I-III

Exclusion Criteria:

* All children with HIV infection attending the HIV clinic at KATH
* Adult HIV patients on ARTs attending the HIV clinic at KATH
* Adult HIV patients with WHO stage IV and V AIDS

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Measure the effects of antimalarials on CD4 cell count decline and HIV viral load increase in study patients | 12 months

SECONDARY OUTCOMES:
Measure the effect of malaria prophylaxis on malaria parasitaemia and haemoglobin levels in study patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Martin-Peprah, MBChB, PhD, Principal Investigator — Komfo Anokye Teaching Hospital
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Kumasi, Ghana